CLINICAL TRIAL: NCT07345130
Title: A Randomized, Open-label, Single-Center, Single-Dose, Three-Treatment, Three-Period, Six-Sequence Crossover Bioequivalence Study of Advil Tablet (Mini) (Ibuprofen 200 mg) to Advil Tablet (Ibuprofen 200 mg) in Healthy Adult Subjects Under Fasted Conditions and Bioavailability Assessment of Advil Tablet (Mini) Under Fed Conditions
Brief Title: A Bioequivalence Study of Advil Tablet (Mini) (Ibuprofen 200 mg) Versus Advil Tablet (Ibuprofen 200 mg) in Healthy Adult Subjects Under Fasted Conditions and Bioavailability Assessment of Advil Tablet (Mini) Under Fed Conditions
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 300286
Record Dates: First submitted 2025-12-12; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Bioequivalence; Bioavailability
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Sequence 1: Treatment A/ Treatment B/ Treatment C (Experimental): Participants will receive a single oral dose of Advil (Mini) tablet under fasted conditions on Day 1 of Period 1 (Treatment A), followed by a single oral dose of Advil tablet under fasted conditions on Day 1 of Period 2 (Treatment B), followed by a single oral dose of Advil (Mini) under fed conditions, on Day 1 of Period 3 (Treatment C). There will be a washout period of at least 3 days between each treatment.
  Interventions: Drug: Advil Tablet (Mini) (Test Product); Drug: Advil Tablet (Reference Product)
- Sequence 2: Treatment B/ Treatment C/ Treatment A (Experimental): Participants will receive a single oral dose of Advil tablet under fasted conditions on Day 1 of Period 1 (Treatment B), followed by a single oral dose of Advil (Mini) under fed conditions, on Day 1 of Period 2 (Treatment C), followed by a single oral dose of Advil (Mini) tablet under fasted conditions on Day 1 of Period 3 (Treatment A). There will be a washout period of at least 3 days between each treatment.
  Interventions: Drug: Advil Tablet (Mini) (Test Product); Drug: Advil Tablet (Reference Product)
- Sequence 3: Treatment C/ Treatment A/ Treatment B (Experimental): Participants will receive a single oral dose of Advil (Mini) under fed conditions, on Day 1 of Period 1 (Treatment C), followed by a single oral dose of Advil (Mini) tablet under fasted conditions on Day 1 of Period 2 (Treatment A), followed by a single oral dose of Advil tablet under fasted conditions on Day 1 of Period 3 (Treatment B). There will be a washout period of at least 3 days between each treatment.
  Interventions: Drug: Advil Tablet (Mini) (Test Product); Drug: Advil Tablet (Reference Product)
- Sequence 4: Treatment A/ Treatment C/ Treatment B (Experimental): Participants will receive a single oral dose of Advil (Mini) tablet under fasted conditions on Day 1 of Period 1 (Treatment A), followed by a single oral dose of Advil (Mini) under fed conditions, on Day 1 of Period 2 (Treatment C), followed by a single oral dose of Advil tablet under fasted conditions on Day 1 of Period 3 (Treatment B). There will be a washout period of at least 3 days between each treatment.
  Interventions: Drug: Advil Tablet (Mini) (Test Product); Drug: Advil Tablet (Reference Product)
- Sequence 5: Treatment B/ Treatment A/ Treatment C (Experimental): Participants will receive a single oral dose of Advil tablet under fasted conditions on Day 1 of Period 1 (Treatment B), followed by a single oral dose of Advil (Mini) tablet under fasted conditions on Day 1 of Period 2 (Treatment A), followed by a single oral dose of Advil (Mini) under fed conditions on Day 1 of Period 3 (Treatment C). There will be a washout period of at least 3 days between each treatment.
  Interventions: Drug: Advil Tablet (Mini) (Test Product); Drug: Advil Tablet (Reference Product)
- Sequence 6: Treatment C/ Treatment B/ Treatment A (Experimental): Participants will receive a single oral dose of Advil (Mini) under fed conditions on Day 1 of Period 1 (Treatment C), followed by a single oral dose of Advil tablet under fasted conditions on Day 1 of Period 2 (Treatment B), followed by a single oral dose of Advil (Mini) tablet under fasted conditions on Day 1 of Period 3 (Treatment A). There will be a washout period of at least 3 days between each treatment.
  Interventions: Drug: Advil Tablet (Mini) (Test Product); Drug: Advil Tablet (Reference Product)

INTERVENTIONS:
Drug: Advil Tablet (Mini) (Test Product) — 200 mg Ibuprofen
Drug: Advil Tablet (Reference Product) — 200 mg Ibuprofen

SUMMARY:
The purpose of this study is to assess the bioequivalence of Advil Tablet (Mini) (Test Product) to Advil Tablet (Reference Product) under fasted conditions and to characterize the impact of food on the bioavailability of the Test Product under fed conditions.

DETAILED DESCRIPTION:
This will be a randomized, open-label, single-center, single-dose, three-treatment, three-period, six sequence crossover bioequivalence and bioavailability (food effect) study in healthy adult participants with at least a 3-day washout period between treatment administrations. A sufficient number of participants will be screened to randomize approximately 50 participants, to ensure that at least 42 evaluable participants complete the entire study. Participants will be randomly assigned to one of six treatment sequences and will receive a single dose of each (of 3) treatments in each (of 3) periods following a crossover design. Blood will be sampled regularly at scheduled times for 24 hours following treatment in each period to assess the pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent form (ICF) indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* A participant whose biological sex at birth is male or female.
* A participant who is 18 to 55 years of age inclusive, at the signing of the ICF.
* A participant who is willing and able to comply with scheduled visits, treatment plan, laboratory tests, study restrictions and other study procedures.
* A participant in good general and mental health with, in the opinion of the Investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon physical examination, vital sign measurements, 12-lead electrocardiogram (ECG) or clinical laboratory tests, or condition, that would impact the participant 's safety, well-being or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* A participant with a body mass index (BMI) of between 18.5 and 30.0 kilogram per meter square (kg/m^2); and a total body weight more than or equal to (>=) 50.0 kg for males and >=45.0 kg for females.
* A female participant of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 30 days after the last dose of assigned treatment. A female participant who is not of childbearing potential must meet at least one of the following criteria:

  1. Has achieved postmenopausal status, defined as cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle-stimulating hormone (FSH) level >=40 milli-international units per milliliter (mIU/mL).
  2. Has undergone a documented (including self-reported) hysterectomy and/or bilateral oophorectomy.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the Investigator; or a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant with, in the opinion of the Investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A female participant who is pregnant (as confirmed by a positive pregnancy test) or intending to become pregnant over the duration of the study.
* A female participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant with any history of asthma, urticaria, or other significant allergic diathesis or allergic reaction to any other pain reliever/fever reducer (example, aspirin or other non-steroidal anti-inflammatory drugs [NSAIDs]). Childhood asthma may be acceptable at the discretion of the Investigator. A participant with uncomplicated seasonal allergic rhinitis can be accepted if expected allergy season is clearly outside enrollment/treatment period.
* A participant with a diagnosis of long QT syndrome or QTcF greater than (>)450 millisecond (msec) for males and >470 msec for females at screening.
* A participant with clinically significant vital sign abnormalities (systolic blood pressure lower than 90 or over 140 millimeter of mercury (mmHg), diastolic blood pressure lower than 50 or over 90 mmHg, or pulse rate less than 50 or over 100 beats per minute [bpm]).
* A participant unwilling or unable to comply with Lifestyle Considerations described in this protocol.
* A participant who has used any medication (including over the counter [OTC] medications and herbal remedies) within 2 weeks or within less than 10 times the elimination half-life of the respective drug (whichever is longer) before first scheduled study drug administration or is anticipated to require any concomitant medication during that period or at any time throughout the study. Allowed treatments are:

  1. systemic contraceptives and hormone replacement therapy, as long as female participant is on stable treatment for at least 3 months before first scheduled study drug administration and continues treatment throughout the study.
  2. occasional use of acetaminophen (up to 2 gram [g] daily).
* A participant with evidence or history of clinically significant laboratory abnormality, hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease within the last 5 years that may increase the risk associated with study participation, in the opinion of the Investigator or medically qualified designee.
* A participant with clinically relevant chronic or acute infectious illnesses or febrile infections within two weeks prior to start of the study.
* A participant who has had any surgical or medical condition which may significantly alter the absorption, distribution, metabolism or excretion of any drug substance.
* A participant with signs and symptoms suggestive of Corona virus disease (COVID)-19 as defined by World Health Organization (WHO) or local guidance (example, fever, cough, etc.) within 14 days prior to the first dose.
* A participant with known COVID-19 positive contacts in the past 14 days.
* A participant who has received any vaccination, including a COVID-19 vaccine, within 14 days prior to the first dose.
* A participant with a history of drug abuse within 1 year prior to screening, or recreational use of soft drugs (such as marijuana) within 1 month, or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to screening.
* A participant with a history of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units for women or 15 units for men of alcohol per week (1 unit = 340 mL of beer 5 percent [%], 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
* A participant with a positive drug screen, alcohol test, or cotinine test.
* A participant who is a current smoker, defined as the use of tobacco or nicotine products during the 3 months prior to screening until admission to the unit or a positive urine cotinine test at screening.
* A participant who reports regular consumption of beverages or food containing xanthine derivatives or xanthine-related compounds (example, coffee, tea, caffeine-containing sodas and chocolate), equivalent to >=500 mg xanthine per day.
* A participant who reports consumption of any drug metabolizing enzyme (example, CYP3A4 or other cytochrome P450 enzymes) inducing or inhibiting aliments, or aliments which have an effect on the P-glycoprotein (PGP) efflux pump (example, beverages or food supplements including broccoli, Brussels sprouts, grapefruit, grapefruit juice, star fruit, pineapple, mango, papaya, St. John's Wort etc.) within 2 weeks prior to admission to the unit.
* A participant with a history of long-term treatment with carbamazepine, phenobarbitone, phenytoin, primidone, rifampicin, St John's Wort or other drugs that induce liver enzymes.
* A participant with positive results in any of the serology tests for human immune deficiency (HIV) antigen and antibody, hepatitis C virus (HCV)-antibody (Ab), hepatitis B serum antigen (HBsAg) and HBc-Ab (immunoglobulin [Ig]G + IgM).
* A participant who has performed strenuous physical exercise (body building, high performance sports) from within 2 weeks prior to admission and who does not agree to refrain from strenuous physical exercise throughout the entire study.
* A participant with an allergy to skin disinfecting agents, tape, or latex rubber, whenever appropriate substitutions cannot be applied or in the Investigator's opinion may pose a risk to the participant.
* A participant with any condition not identified in the protocol that in the opinion of the Investigator would confound the evaluation and interpretation of the study data or may put the participant at risk.
* A participant who has donated plasma within 7 days prior to first dosing, or who has donated or lost 500 mL or more of whole blood within 8 weeks prior to first dosing.
* A participant with veins unsuitable for repeated venipuncture, as assessed at screening by the Investigator or suitably qualified designee.
* A participant who, in the opinion of the Investigator or medically qualified designee, should not participate in the study.
* A participant who has previously been enrolled in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Post-dose Concentration (Cmax) Under Fasted Conditions (Test Versus (vs) Reference Product) | Pre-dose (within 1 hour prior to dosing) and at 5,10,15,30,45 minutes and 1,1.25,1.5,1.75,2,2.25,2.5,2.75,3,3.25,3.5,3.75,4,4.25,4.5,4.75,5,5.5,6,8,10,12,16 and 24 hours post-dose on Day 1 in each treatment period (each treatment period is 3 days)
  Cmax is defined as the maximum observed post-dose concentration obtained without interpolation. Blood samples will be collected at indicated timepoints for the analysis of Cmax.
Area Under the Plasma Concentration Versus Time Curve Calculated from Time 0 to the Last Measurable Sampling Time Point, t (AUC[0-t]) Under Fasted Conditions (Test Vs Reference Product) | Pre-dose (within 1 hour prior to dosing) and at 5,10,15,30,45 minutes and 1,1.25,1.5,1.75,2,2.25,2.5,2.75,3,3.25,3.5,3.75,4,4.25,4.5,4.75,5,5.5,6,8,10,12,16 and 24 hours post-dose on Day 1 in each treatment period (each treatment period is 3 days)
  AUC(0-t) is defined as the area under the plasma concentration versus time curve calculated from time 0 to the last measurable sampling time point, t, computed using the linear trapezoidal rule. Blood samples will be collected at indicated timepoints for the analysis of AUC(0-t).
Cmax for Test Product Under Fed Conditions Compared to Fasted Conditions | Pre-dose (within 1 hour prior to dosing) and at 5,10,15,30,45 minutes and 1,1.25,1.5,1.75,2,2.25,2.5,2.75,3,3.25,3.5,3.75,4,4.25,4.5,4.75,5,5.5,6,8,10,12,16 and 24 hours post-dose on Day 1 in each treatment period (each treatment period is 3 days)
  Cmax is defined as the maximum observed post-dose concentration obtained without interpolation. Blood samples will be collected at indicated timepoints for the analysis of Cmax.
AUC(0-t) for Test Product Under Fed Conditions Compared to Fasted Conditions | Pre-dose (within 1 hour prior to dosing) and at 5,10,15,30,45 minutes and 1,1.25,1.5,1.75,2,2.25,2.5,2.75,3,3.25,3.5,3.75,4,4.25,4.5,4.75,5,5.5,6,8,10,12,16 and 24 hours post-dose on Day 1 in each treatment period (each treatment period is 3 days)
  AUC(0-t) is defined as the area under the plasma concentration versus time curve calculated from time 0 to the last measurable sampling time point, t, computed using the linear trapezoidal rule. Blood samples will be collected at indicated timepoints for the analysis of AUC(0-t).
Area Under the Plasma Concentration Versus Time Curve Calculated From Time 0 to Infinity (AUC[0-inf]) for Test Product Under Fed Conditions Compared to Fasted Conditions | Pre-dose (within 1 hour prior to dosing) and at 5,10,15,30,45 minutes and 1,1.25,1.5,1.75,2,2.25,2.5,2.75,3,3.25,3.5,3.75,4,4.25,4.5,4.75,5,5.5,6,8,10,12,16 and 24 hours post-dose on Day 1 in each treatment period (each treatment period is 3 days)
  AUC(0-inf) is defined as the area under the plasma concentration versus time curve calculated from time 0 to infinity. AUC(0-inf) = AUC(0-t) + C(t)/λz where C(t) is the concentration at the last measurable sampling time point and λz is the terminal elimination rate constant. Blood samples will be collected at indicated timepoints for the analysis of AUC(0-inf).

SECONDARY OUTCOMES:
AUC(0-inf) for Test and Reference Products | Pre-dose (within 1 hour prior to dosing) and at 5,10,15,30,45 minutes and 1,1.25,1.5,1.75,2,2.25,2.5,2.75,3,3.25,3.5,3.75,4,4.25,4.5,4.75,5,5.5,6,8,10,12,16 and 24 hours post-dose on Day 1 in each treatment period (each treatment period is 3 days)
  AUC(0-inf) is defined as the area under the plasma concentration versus time curve calculated from time 0 to infinity. AUC(0-inf) = AUC(0-t) + C(t)/λz where C(t) is the concentration at the last measurable sampling time point and λz is the terminal elimination rate constant. Blood samples will be collected at indicated timepoints for the analysis of AUC(0-inf).
Percentage of AUC(0-inf) Obtained by Extrapolation (%AUCex) for Test and Reference Products | Pre-dose (within 1 hour prior to dosing) and at 5,10,15,30,45 minutes and 1,1.25,1.5,1.75,2,2.25,2.5,2.75,3,3.25,3.5,3.75,4,4.25,4.5,4.75,5,5.5,6,8,10,12,16 and 24 hours post-dose on Day 1 in each treatment period (each treatment period is 3 days)
  %AUCex is defined as the percentage of AUC(0-inf) obtained by extrapolation, calculated as (1-[AUC0-t/AUC0-inf]) *100. Blood samples will be collected at indicated timepoints for the analysis of %AUCex.
Terminal Elimination Rate Constant (λz) for Test and Reference Products | Pre-dose (within 1 hour prior to dosing) and at 5,10,15,30,45 minutes and 1,1.25,1.5,1.75,2,2.25,2.5,2.75,3,3.25,3.5,3.75,4,4.25,4.5,4.75,5,5.5,6,8,10,12,16 and 24 hours post-dose on Day 1 in each treatment period (each treatment period is 3 days)
  λz is defined as the terminal elimination rate constant computed as the negative of the slope of the regression line of ln(C[t]) on time. The regression should generally involve at least 3 consecutive measurable concentrations that decrease over time excluding Cmax. Blood samples will be collected at indicated timepoints for the analysis of λz.
Time of the Maximum Observed Post-dose Concentration (tmax) for Test and Reference Products | Pre-dose (within 1 hour prior to dosing) and at 5,10,15,30,45 minutes and 1,1.25,1.5,1.75,2,2.25,2.5,2.75,3,3.25,3.5,3.75,4,4.25,4.5,4.75,5,5.5,6,8,10,12,16 and 24 hours post-dose on Day 1 in each treatment period (each treatment period is 3 days)
  Blood samples will be collected at indicated timepoints for the analysis of tmax.
Elimination Half-life (t1/2) for Test and Reference Products | Pre-dose (within 1 hour prior to dosing) and at 5,10,15,30,45 minutes and 1,1.25,1.5,1.75,2,2.25,2.5,2.75,3,3.25,3.5,3.75,4,4.25,4.5,4.75,5,5.5,6,8,10,12,16 and 24 hours post-dose on Day 1 in each treatment period (each treatment period is 3 days)
  t1/2 is defined as the elimination half-life computed as t1/2 = ln(2)/λz where λz is the terminal elimination rate constant. Blood samples will be collected at indicated timepoints for the analysis of t1/2.
Apparent Volume of Distribution (Vz/F) for Test and Reference Products | Pre-dose (within 1 hour prior to dosing) and at 5,10,15,30,45 minutes and 1,1.25,1.5,1.75,2,2.25,2.5,2.75,3,3.25,3.5,3.75,4,4.25,4.5,4.75,5,5.5,6,8,10,12,16 and 24 hours post-dose on Day 1 in each treatment period (each treatment period is 3 days)
  Vz/F is defined as the apparent volume of distribution, as calculated by the dose administered/(λz *AUC0-inf) where λz is the terminal elimination rate constant and AUC(0-inf) is the area under the plasma concentration versus time curve calculated from time 0 to infinity. Blood samples will be collected at indicated timepoints for the analysis of Vz/F.
Apparent Total Clearance (Cl/F) for Test and Reference Products | Pre-dose (within 1 hour prior to dosing) and at 5,10,15,30,45 minutes and 1,1.25,1.5,1.75,2,2.25,2.5,2.75,3,3.25,3.5,3.75,4,4.25,4.5,4.75,5,5.5,6,8,10,12,16 and 24 hours post-dose on Day 1 in each treatment period (each treatment period is 3 days)
  Cl/F is defined as the apparent total clearance, as calculated by the dose administered/AUC0-inf where AUC(0-inf) is the area under the plasma concentration versus time curve calculated from time 0 to infinity. Blood samples will be collected at indicated timepoints for the analysis of Cl/F.
Number of Participants Reporting Ease of Swallowing: Categorical Response | Post Dose on Day 1 in each treatment period (each treatment period is 3 days)
  Immediately after dosing, participants will be asked to evaluate the ease of swallowing to assess the acceptability of each treatment. Participants will be asked to provide a categorical response (Agree/Disagree) to the question "Do you agree or disagree that the product is easy to swallow?".
Number of Participants Reporting Ease of Swallowing on a 5-Point Ordinal Scale | Post Dose on Day 1 in each treatment period (each treatment period is 3 days)
  Immediately after dosing, participants will be asked to rank the ease of swallowing of each product on a 5-point ordinal scale with scores ranging from 1 to 5 where 1=not easy to swallow; 2=somewhat easy to swallow; 3=average to swallow; 4=above average to swallow; 5=very easy to swallow. Higher score indicates more ease in swallowing.

CONTACTS AND LOCATIONS:
Locations (1):
- Novum Pharmaceutical Research Services, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.